CLINICAL TRIAL: NCT04758611
Title: Pilot Study to Evaluate the Safety and Effectiveness of the CereVasc eShunt™ System in the Treatment of Communicating Hydrocephalus
Brief Title: The ETCHES I Study (Endovascular Treatment of Communicating Hydrocephalus With an Endovascular Shunt)
Acronym: ETCHES I
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CereVasc Inc (Industry)
Collaborators: AlvaMed, Inc. (Industry); Bioscience Consulting, Inc. (Industry); Simplified Clinical Data Systems, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN-0001
Record Dates: First submitted 2021-02-09; First posted 2021-02-17 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Hydrocephalus, Communicating; Hydrocephalus
Keywords: eShunt
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Intervention Model Description: Prospective, single-center, open-label, single-arm pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Treatment Arm (Experimental): The Treatment Arm receives the eShunt implant
  Interventions: Device: eShunt™ Implant

INTERVENTIONS:
Device: eShunt™ Implant — The eShunt™ Implant is designed to drain excess cerebrospinal fluid (CSF) from the intracranial subarachnoid space (SAS) into the venous system as a minimally invasive treatment for communicating hydrocephalus.
  Other Names: eShunt™; eShunt™ System

SUMMARY:
The eShunt™ System is a minimally invasive method of treating communicating hydrocephalus. The eShunt System includes a proprietary eShunt Delivery System and the eShunt Implant, a permanent implant deployed in a minimally invasive, neuro-interventional procedure. The eShunt Implant is designed to drain excess cerebrospinal fluid (CSF) from the intracranial subarachnoid space (SAS) into the venous system.

DETAILED DESCRIPTION:
This is a prospective, single-center, open label, single-arm pilot study of the eShunt System. The study population consists of patients with post-aneurysmal subarachnoid hemorrhage (SAH) treated for increased intracranial pressure (ICP) resulting in symptomatic hydrocephalus using an external ventricular drain (EVD) to facilitate CSF drainage and who cannot be "weaned" from the EVD following the hemorrhagic event.

The study will be performed a single site with up to 30 subjects who meet the inclusion and exclusion criteria for the study. Subjects will be evaluated every 30 days for the first 90 days following eShunt Implant deployment with standard neurological evaluation appropriate for patients with communicating hydrocephalus. In addition, follow-up will occur at 180 days, 12 and 24 months post-operatively and will include imaging in addition to the standard neurological evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18
2. Subject provides Informed Consent (IC)
3. Post-aneurysmal SAH with Hunt and Hess Grades I-IV with EVD in place with the need for a permanent CSF shunt determined through a failed EVD clamping trial defined as:

   1. Post-clamping ICP of > 20 cmH2O for 15 min, or
   2. Post-clamping ICP > 25 cmH2O for < 15 min with patient intolerance to EVD clamping
   3. Post-clamping ICP >15 cmH2O for 15 min with radiographic evidence of ventriculomegaly
4. Clinical signs and symptoms of communicating hydrocephalus
5. Neurologically stable without evidence of severe vasospasm
6. Pre-procedure MRI with gadolinium confirmation of IPS (inferior petrosal sinus) and CPA (cerebellopontine angle) cistern anatomy suitable for eShunt Implant deployment as confirmed by SSC (subject screening committee)
7. Pre-procedure CT confirmation of no obstruction preventing CPA cistern access at target implant site (e.g., petrous bone) as confirmed by SSC

Exclusion Criteria:

1. Patient is in a state of unconsciousness or is unable to understand the information provided in the Informed Consent Form for this study
2. Indication of obstructive hydrocephalus
3. Presence of gross blood in CSF from EVD
4. Pregnant
5. Unwilling or unable to comply with follow up requirements
6. Active systemic infection or infection detected in CSF
7. Life expectancy < 1 year
8. Hypersensitivity or contraindication to heparin or radiographic contrast agents which cannot be adequately pre-medicated, desensitized or where no alternative is available
9. Occlusion or stenosis of the internal jugular vein
10. Venous distension in the neck on physical exam
11. Atrial septal defect or patent foramen ovale identified on cardiac echocardiogram
12. History of bleeding diatheses, coagulopathy or will refuse blood transfusion in cases of emergency
13. Clearly antecedent stroke unrelated to post-aneurysmal SAH
14. Patient is currently participating in another investigational drug or device trial that could conflict with study data collection or follow-up
15. Other medical illnesses that may cause the patient to be non-compliant with the protocol or confound data interpretation as determined by the study Investigator
16. Presence of a deep vein thrombosis superior to the popliteal segment of the femoral vein
17. International Normalized Ratio (INR) or Partial Thromboplastin Time (PTT) results outside of normal range (INR 0.8-1.4; PTT 25-35 secs.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in intracranial pressure (ICP) | 36-48 hours following eShunt Implant deployment
  At 36-48 hours following eShunt Implant deployment and with EVD remaining clamped, an ICP assessment that demonstrates: 1) ICP below 20 cmH2O as measured by the EVD with no periods longer than 15 minutes above 20 cmH2O; and 2) No episodes of ICP, measured by EVD, above 25 cmH2O with associated subject symptoms

SECONDARY OUTCOMES:
Number of subjects requiring conversion to conventional CSF shunt | 24 months following eShunt Implant deployment
  Evaluate the need for CSF diversion by conventional CSF shunt insertion within the 24 months following eShunt Implant deployment
Incidence of clinically significant abnormal laboratory test results | 24 months following eShunt Implant deployment
  Clinically significant changes from baseline laboratory test results will be summarized
Incidence of clinically significant changes from baseline MRI imaging | 24 months following eShunt Implant deployment
  Clinically significant changes from baseline MRI images will be summarized
Incidence of clinically significant changes from baseline CT imaging | 24 months following eShunt Implant deployment
  Clinically significant changes from baseline CT images will be summarized

OTHER OUTCOMES:
Safety Endpoint: serious adverse events (SAEs) | 24 months following eShunt Implant deployment
  Evaluate for any device or procedure related serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Pedro M Lylyk, MD, Principal Investigator — Clinica Sagrada Familia
Locations (1):
- Clínica La Sagrada Familia, Buenos Aires, Ciudad A. de Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heilman CB, Basil GW, Beneduce BM, Malek AM. Anatomical characterization of the inferior petrosal sinus and adjacent cerebellopontine angle cistern for development of an endovascular transdural cerebrospinal fluid shunt. J Neurointerv Surg. 2019 Jun;11(6):598-602. doi: 10.1136/neurintsurg-2018-014445. Epub 2019 Jan 9. PMID 30626626
- [Result] Lylyk P, Lylyk I, Bleise C, Scrivano E, Lylyk PN, Beneduce B, Heilman CB, Malek AM. First-in-human endovascular treatment of hydrocephalus with a miniature biomimetic transdural shunt. J Neurointerv Surg. 2022 May;14(5):495-9. doi: 10.1136/neurintsurg-2021-018136. Epub 2021 Dec 3. PMID 34862267
- [Derived] Amllay A, Matouk CC. A Paradigm Shift in Hydrocephalus Management: The Promise of Endovascular Cerebrospinal Fluid Diversion. Cardiol Rev. 2025 Jul-Aug 01;33(4):294-297. doi: 10.1097/CRD.0000000000000886. Epub 2025 Mar 26. PMID 40135887